CLINICAL TRIAL: NCT02263222
Title: A Feasibility Dose-escalating Study to Evaluate the Tolerability and Systemic Exposure of MDT-10013 Plus Routine Care in the Treatment of Acute Postoperative Pain Following Total Knee Arthroplasty
Brief Title: A Feasibility Dose-escalating Study of MDT-10013 for Acute Postoperative Pain Following Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P13-02
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Post-operation Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDT-10013 (Experimental): Subjects will receive MDT-10013.
  Interventions: Drug: MDT-10013

INTERVENTIONS:
Drug: MDT-10013

SUMMARY:
This is an open-label dose-escalating study to evaluate the tolerability and systemic exposure of MDT-10013 in men and women at least 18 years of age who are undergoing primary unilateral TKA.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female at least 18 years of age
2. Has a body mass index from 18 kg/m2 to 40 kg/m2
3. Is scheduled to undergo standard primary (first-time) unilateral TKA surgery (due to osteoarthritis) with or without patellar resurfacing. Standard conventional instrumentation and cemented components must be used and the surgery shall be conducted under spinal anesthesia.
4. Females must meet the following criteria:

   * Is of nonchildbearing potential, defined as any woman who has undergone surgical sterilization or is more than 2 years postmenopausal
   * If of childbearing potential, may be enrolled if pregnancy test results are negative at Screening and if she is routinely using an effective method of birth control with a low failure rate (i.e., hormonal contraception, intrauterine device, condoms in combination with a spermicidal cream, or total sexual abstinence).
   * May not be pregnant or lactating
5. Has read, understood, and signed the informed consent before study entry
6. Is mentally competent, reliable, and cooperative to undergo all visits and procedures scheduled in the study protocol and to record the required information.

Exclusion Criteria:

1. Has had previous spinal surgery or other contraindications that preclude use of spinal anesthesia or is not indicated for surgery because of an inflammatory process or risk of infection or delayed wound healing (e.g., autoimmune disorder)
2. Is scheduled to undergo a concurrent surgical procedure (e.g., bilateral TKA)
3. Has a concurrent painful condition or surgery that may require analgesic treatment (such as a nonsteroidal antiinflammatory drug [NSAID] or opioid) in the postsurgical period for pain not strictly related to the TKA, and that may confound postsurgical assessments
4. Has a history of allergy or hypersensitivity to the components in the investigational product or to the routine care medications
5. Has current orthostatic hypotension (i.e., systolic blood pressure decrease of at least 20 mmHg or diastolic blood pressure decrease of at least 10 mmHg or an increase in heart rate of 20 beats per minute within 3 minutes of standing)
6. Has any clinically significant cardiovascular condition as evidenced by physical examination, medical history, and/or baseline electrocardiogram (ECG), including inadequately controlled hypertension
7. Has evidence of bradycardia as shown by heart rate of <50 beats per minute via screening ECG
8. In the investigator's opinion, subject is not a suitable candidate for study treatment and/or has any poorly controlled or serious medical conditions, psychiatric illnesses, or clinically significant laboratory values that the investigator suspects could compromise the subject's safety or the scientific integrity of the study (e.g., human immunodeficiency virus [HIV], hepatitis B or C [hep B, hep C])
9. Has presence or history of local or systemic malignant disease in the past 5 years (history of basal cell carcinoma will be allowed)
10. Has undergone prior open surgery in the affected knee
11. Has impaired renal function (creatinine >1.5 times upper limit of normal)
12. Has chronic liver function impairment (aspartate aminotransferase or alanine aminotransferase >3 times upper limit of normal)
13. Has insulin-dependent diabetes or uncontrolled diabetes mellitus (glycosylated hemoglobin >7%)
14. Has leukopenia (<3500 leukocytes/μL)
15. Has current treatment with any of the following medications:

    1. Systemic corticosteroids within 1 month of the planned surgery (intranasal/inhaled steroids are acceptable)
    2. Immunosuppressant therapy to treat autoimmune diseases (e.g., rheumatoid arthritis, multiple sclerosis, myasthenia gravis, systemic lupus erythematosus, sarcoidosis, focal segmental glomerulosclerosis, Crohn's disease, Behcet's disease, pemphigus, or ulcerative colitis)
    3. Oral or topical products containing clonidine (e.g., Catapres®)
    4. Antiepileptic drugs, antipsychotics, monoamine oxidase inhibitors, lithium, or sulfonamides
    5. Calcium channel blocker, digoxin, or beta-adrenergic blockers
16. Chronically uses opioids, defined as use on at least 20 of the last 30 days before study Screening, and is unable to refrain from opioid use within the 24 hour period before surgery
17. Investigator determines subject has a known or suspected history of drug or alcohol abuse
18. Recent dose adjustment or commencement of treatment with selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), and/or tricyclic antidepressants (use of these medications is allowed if the dose is stable for at least 8 weeks before receiving study treatment)
19. Has received any other investigational drug or device within 30 days of Screening
20. Experiences any surgical complication that, in the investigator's opinion, precludes implantation of MDT-10013.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters of MDT-10013--maximum plasma concentration observed (Cmax) | From day 1 to day 14
Pharmacokinetic (PK) parameters of MDT-10013--time to maximum plasma concentration observed (tmax) | From day 1 to day 14
Pharmacokinetic (PK) parameters of MDT-10013--area under the plasma concentration versus time curve (AUC) | From day 1 to day 14
Rate of study drug/treatment-related serious adverse events (SAEs) | up to 3 months

SECONDARY OUTCOMES:
Summed pain intensity scores at rest | up to 120 hours
  Summed pain intensity scores (calculated as a time-weighted average) by using an 11-point (0 to 10) numerical rating scale (NRS).
Summed pain intensity scores over 2 to 48 hours (SPI-48) with activity | up to 48 hours
Aggregate dosage of all opioid analgesia | 0 to 24 hours and 0 to 48 hours
Total use of opioid analgesia | From 48 hours through Day 6/120 hours
Time to first use of opioid analgesia defined as the time from Time 0 to the first use of opioid analgesia. | Time 0 is defined as the initiation of arthrotomy closure to the first opioid analgesia use
Subject global evaluation of study treatment | up to 10-14 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Florida Research Associates, LLC, DeLand, Florida
  - Clinical Research Department, University of Orthopedics Center, Altoona, Pennsylvania